CLINICAL TRIAL: NCT00206778
Title: A Randomized Open-Label 6 Month Acute and Maintenance Trial of Lamotrigine vs. Standard of Care Sodium Valproate Monotherapy for Treatment of Mixed Mania.
Brief Title: Six Month Trial of Lamotrigine vs. Sodium Valproate for Treatment of Mixed Mania
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Igor Galynker, MD, Beth Israel Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 100-03
Record Dates: First submitted 2005-09-16; First posted 2005-09-21 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-11

CONDITIONS: Mixed Mania Bipolar Disorder
Keywords: Mixed mania; Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lamotrigine; Valproic Acid

INTERVENTIONS:
Drug: Lamotrigine
Drug: Sodium Valproate

SUMMARY:
We are comparing the efficacy of Lamotrigine to that of Standard of Care Sodium Valproate for the treatment of Mixed Mania. The study hypothesis is that Lamotrigine will be more efficative for treating mixed mania in patients with Bipolar Disorder.

DETAILED DESCRIPTION:
Mixed mania is a clinically distinct affective state which is likely to be more severe than classical euphoric mania and to have longer episode duration. Mixed mania is associated with longer duration of illness, suicidality, and poor outcome (McElroy et al, 1995). Although at present there is no universally agreed on definition for mixed states, 40-60% of patients in acute manic states also meet criteria for either major depression or dysphoria (Dilsaver et al,1999; Calabrese et al, 1999; Secunda et al,1985; Sporn and Sacks,1997). Dilsaver at al (1999) in their factor analytic study of manic symptoms were able to differentiate dysphoric and depressed mania. Patients with depressed mania (30% of all patients with mania) were as manic as patients with euphoric mania and also met criteria for the Major depressive disorder. Patients with dysphoric mania were less manic and less depressed, but more irritable than both depressed and euphoric manic patients.

At present there is no accepted treatment algorithms for mixed affective states including depressed and dysphoric mania in Dilsaver definition. Currently used antimanic agents (lorazepam, typical antipsychotics, olanzapine) and mood stablizers (lithium, divlaproex sodium) have little or no antidepressant activity. Therefore, treatment of mixed mania frequently results in emergence of bipolar depression that is often treatment-refractory. Thus is an urgent need for effective treatment of mixed mania that will not result in bipolar depression.

Lamotrigine is an anticonvulsant that prolongs the refractory phase of voltage sensitive channels, an action that is associated with antimanic properties (Hurly, 2002; Sporn and Sacks, 1997; Calabrese et al; 1999, Normann et al; 2002). Lamotrigine was postulated to decrease glutamate release by acting at voltage-sensitive sodium channel in their refractory phase, stabilizing presynaptic neuronal membranes and inhibiting pathologic release of glutamate. As abnormalities in glutamatergic system have been implicated in depression, and NMDA receptor antagonists reverse anxiety or depression in various stress models, lamotrigine could act as an antidepressant. . Thus, lamotrigine has a potential to have both antimanic and antidepressant activity (for refs, see Sporn and Sacks, 1997), and in theory should be uniquely effective for mixed mania (Dilsaver et al, 1999). Indeed, clinical trials reviewed in detail by Hurley (2002), demonstrated that lamotrigine is somewhat effective an antimanic agent, and has significant antidepressant activity in bipolar depression. Lamotrigine was used in a combination with other agents or as monotherapy, and the response rates for depressed, mixed and rapid cycling states were similar, ranging from 52% to 63%. With slow dose titration (6 weeks), side effects were few and the incidence of exfoliative dermatitis was 1 in 500. Of note, although Sporn and Sachs (1997) reported a switch from depression to rapid cycling, such incidences were few. In our institution, lamotrigine was effective for treatment of mixed mania and bipolar depression in patients receiving standard maintenance treatment for Bipolar Mood Disorder. Lamotrigine did worsen agitation in two elderly patients with symptoms of irritable mania.

Based on the above evidence, it appears that lamotrigine, either in combination with a proven antimanic agent or in monotherapy, is uniquely suited to be the agent of choice for treatment of mixed mania. Therefore, we here propose a randomized open-label trial of lamotrigine vs. standard of care sodium valpoate for treatment of mixed mania. Within this framework, the following are the study's hypotheses and objectives:

Hypothesis/Objectives Objective One. To compare the efficacy of the lamotrigine with sodium valproate (standard of care) for treatment of depressive symptoms of acute mania in patients with Bipolar Mood Disorder.

Hypothesis One:

Lamotrigine will be more effective than sodium valproate in treatment of depressive symptoms in acute mixed mania.

Objective Two. To compare the efficacy of the lamotrigine with that of sodium valproate for treatment of manic symptoms in acute mixed mania.

Hypothesis Two:

Lamotrigine and sodium valproate will be equally effective in treatment of manic symptoms in acute mixed mania as measured by the Young Mania Rating Scale scores.

Objective Three. To compare the efficacy of lamotrigine to that of sodium valproate in maintenance treatment of patients with bipolar mood disorder and a recent past episode of mixed mania.

Hypothesis Three:

(i)The lamlotrigine will be more efficacious than sodium valproate in maintenance treatment of patients with bipolar mood disorder and a recent past episode of mixed mania.

(ii) The lamotrigine patients will have lower relapse rate. (iii) The lamotrigine patients will have lower rates of depression than patients treated with sodium valproate.

Objective Four: To compare the side effect profile of lamotrigine treatment of mixed mania to sodium valproate treatment of mixed mania in patients with bipolar mood disorder and a recent past episode of mixed mania.

Hypothesis four:

Lamotrigine acute treatment will result in comparable side effect profile with that of sodium valproate while lamotrigine maintenance treatment will be superior to that with sodium valproate.

Methods We plan to study two eighteen-subject groups (36 subjects total) of male and female study participants between ages 18 and 65 over a 1 1/2 year period. The subjects will be enrolled from the inpatient units at the Beth Israel Medical Center and at the St. Lukes-Roosevelt Hospital Center (Continuum Health Partners) and will be followed at the Center for Treatment of the Affective Disorders in the Department of Psychiatry at BIMC. An independent evaluator (Paul Teusink, M.D.) not affiliated with the study will determine capacity of consent. We will select patients who would have had at least one prior manic episode and who meet inclusion and exclusion criteria for depressed acute mania (Dilsaver et al, 1999). The study criteria for an acute episode of irritable depressed mania will be a Young Mania Rating Scale (YMRS) score of at least 11 and the Hamilton Depression Rating Scale (HDRS) score of at least 18 with 72 hours prior to entering the study. Patient could be randomized on study medication if she/he came to clinic on lamotrigine or Sodium valprole, but she/he has low blood level of this drug.

The study will have two phases.

Phase 1, The Acute Phase. Index medications schedule. Following randomization, during the first 8-week phase, the index manic episode will be treated with either adjust lamotrigine or sodium valproate will be started at 25 mg po daily and will be increased biweekly until a maximal dose of 200 mg/day. Dose escalation schedule: weeks 1-2 25 mg po qd, week 3-4 25 mg po bid, weeks 5-6 50 mg po bid, weeks 7-8 100 mg po bid. The dose could be decreased to as low as 50 mg/day to reduce side effects other than rash. The sodium valproate treatment will be initiated with a loading dose of 20 mg/kg, and the dose will be adjusted in 250 mg/day increments to achieve a therapeutic level of 100-120 mcg/kg.

Concomitant medications schedule. If a patient is receiving mood stabilizers such as lithium, , carbamazepine, gabapentine, trileptal, lamotrigine or sodium valproate at the beginning of the study, these medications will be discontinued in 72 hours informed consent is provided. The following medications will not be permitted during the acute phase of the trial: clozaril, depot neuroleptics antipsychotic, antidepressant and benzodiazepines other than lorazepam.

Rescue medications. Since neuroleptics and lorazepam will be liberally allowed for treatment of acute manic symptoms, no rescue medications will be necessary in the acute phase.

Crossover design for subjects with treatment failure. If subject's condition deteriorates after randomization to lamotrigine or valporate, subject will be crossed over to the other arm of the study, i.e. those who failed sodium valproate will be treated with lamotrigine and vise versa and vise versa. Subjects who will have failed the crossover switch will be removed from the study. Deterioration will be defined as a three-point worsening in the patient's YMRS score lasting more than 72 hours.

Outcome measures. The severity of illness will be measured with Young Mania Rating Scale (MRS), Hamilton Rating scale for depression, and the CGI rating scale. The primary outcome measures will be the YMRS total score change from baseline until the endpoint of Phase 1. The secondary outcome measures will be the HRSD total score change and the CGI score change from baseline until the Phase 1 endpoint. Other secondary outcome measures will be the amount the incidences of seclusion and restraint, the length of hospital stay, and the medical indeces such as HgA1C, weight changes, and lipid profile

Phase 2, The Maintenance Phase. If after two month of treatment patient improve on 50% compare to initial level of YMRS , HDRS and YMRS<11, HDRS<18 patient will be transferred to the Maintenance Phase. Index Medication Schedule.

The acute phase will be followed by the 4 months maintenance phase. In the maintenance phase, all medications but lorazepam (< 4 mg/ day dose) and lamotrigine or sodium valproate will be typed over for initial 4 weeks period. In the last 3 month of the study the lamotrigine subjects will receive only lamotrigine monotherapy. The dose will be adjusted by the study physicians as clinically necessary within the same dose range as in the Phase 1. The sodium valproate dose will be maintained to achieve a therapeutic level of 50-100 mcg/ml. The subjects will be followed weekly for the first 5 weeks of the study. For the rest of the study the subjects will be followed biweekly

Rescue medications schedule. During the maintenance phase, lorazepam will be tapered to a minimal dose that would allow nightly sleep of at least 8 hrs. The dose adjustment will be done weekly according to the following dose reduction schedule: 4 mg - 3 mg - 2 mg - 1 mg - 0 5 mg - 0 mg and will take up to five weeks depending on the initial dose.

Outcome measures. The primary outcome measures will be the number and the time to either manic or depressive episodes. The secondary outcome measures will be an average change from baseline in YMRS, HRSD, and CGI scores from baseline until the endpoint of Phase 2. We will also evaluate medication side effects, the need for adjunct lorazepam treatment, the reasons for premature discontinuation, the demographic data, and the medical endpoints (HgbA1C, weight changes, lipid profile). We will use SPSS and appropriate statistical methods for statistical analysis.

Study Population

The patient population will consist of psychiatric inpatients at the Beth Israel Medical Center and the St. Lukes-Roosevelt Hospital Center, who meet criteria for the DSM-IV diagnosis of Bipolar Mood Disorder I, manic episode. At present, the patient ethnic and racial mix is 26% Hispanic, 30% African American, and 45% Caucasian. The gender distribution is 46% male, 54% female. The inpatient payer mix is 26% Medicare and 50% Medicaid. The average length of stay for the three units is 19 days for all patients and 26 days for patients without co-morbid substance use.

In 1999-2001, inpatient units at the BIMC registered on average 1500 yearly admissions, 1350 of them ages 17-65. Upon admission, approximately 200 patients carried a diagnosis of Bipolar Mood Disorder I, manic episode, without comorbid substance abuse. The inpatient units at Saint Lukes Roosevelt admit 100 manic patients yearly. If the admission demographics remain unchanged for 2003, we expect that 40 patients per year will meet diagnostic inclusion criterion for the study. Based on our previous experience with recruitment for research studies, we expect that 30 % of patients meeting the diagnostic criteria will also meet other inclusion and exclusion criteria, will sign the inform consent and participate in the study. Therefore we expect to recruit 36 patients per year and to complete the study accrual in 18 months. We plan to complete the data analysis for the acute phase within one year.

Inclusion Criteria

1. Males and females, ages 18-65.
2. Ability to sign an informed consent
3. Diagnosis of Bipolar Mood Disorder I, manic episode.
4. Mania Rating Scale (MRS) score of at least 11
5. HDRS score of at least 18
6. Global Assessment Scale (GAS) scores more than 60. Exclusion Criteria

1) Alcohol or substance abuse within the last 6 months 2) Current diagnosis of Obsessive-Compulsive Disorder 3) Current diagnosis of Schizophrenia or Schizoaffective Disorder 4) Previous adverse reaction or allergies to lamotrigine or sodium valproate

Study Design and Drug Regimens The study will be months open label parallel comparison (with a blinded rater) of combination therapy lamotrigine 25-200 mg/day(flexible dosing) and sodium valproate (flexible dosing) monotherapy for treatment of mixed mania in two groups of patients with Bipolar Mood Disorder I. The study will have acute and maintenance phases. Each group will consist of 18 subjects matched for age, gender, and education.

Data Analysis

All patients who were randomly assigned to treatment groups and had at least one post-baseline assessment will be included in the efficacy analysis. The primary time points will be the endpoints of Phases 1 and 2 (i.e. the last available observation during Phases 1 and 2). The primary comparison will be between the lamotrigine/ sodium valproate groups. The analysis of covariance model will be used to test differences between treatments at endpoint. The model will include factors for treatment, and baseline scores on MRS and HRDS as a covariate. MRS scores at all time points will be analyzed jointly by means of repeated measures model. HRDS scores will be analyzed in the same way as MRS scores. Treatment over time will be used as a factor in the model. Gehan's generalized Wilcoxon test will be used to evaluate differences in time to discontinuation (ref from Sachs), and Van Elteren test will be used to evaluate differences in the CGI scores (ref from Sachs).

Scientific Relevance and Health Implications

The successful completion of this study will indicate that lamotrigine combination should be the preferred first-line treatment for mixed mania that should be continued as the preferred maintenance treatment for mixed mania.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ages 18-65.
* Ability to sign an informed consent
* Diagnosis of Bipolar Mood Disorder I, manic episode.
* Mania Rating Scale (MRS) score of at least 11
* HDRS score of at least 18
* Global Assessment Scale (GAS) scores more than 60.

Exclusion Criteria:

* Alcohol or substance abuse within the last 6 months
* Current diagnosis of Obsessive-Compulsive Disorder
* Current diagnosis of Schizophrenia or Schizoaffective Disorder
* Previous adverse reaction or allergies to lamotrigine or sodium valproate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2003-07; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Igor Galynker, MD, PhD, Principal Investigator — Beth Israel Medical Center
Locations (1):
- Beth Israel Medical Center, New York, New York, United States